CLINICAL TRIAL: NCT06483100
Title: Measurable Residual Disease-Guided Post-Transplant Elranatamab Maintenance
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Comprehensive Cancer Network (Network); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202409141
Record Dates: First submitted 2024-06-25; First posted 2024-07-03 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma
Keywords: Maintenance; Stem cell transplant; Immunotherapy
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Elranatamab (Experimental): Patients will receive at least 12 months of maintenance elranatamab therapy. Patients will have MRD testing within clonoSEQ every 6 months. If 2 consecutive tests are negative, elranatamab will be stopped and the patient will go on observation schedule.
  Once a patient starts the observation schedule, standard disease monitoring will be performed every 3 months and bone marrow-based MRD will be performed every 6 months until MRD recurrence, disease progression or end of study period (patients' on-study status will be a maximum of 36 months for treatment and intensive observation combined). Patients who experience MRD recurrence will be re-treated per study protocol. A patient may move back to the observation schedule after treatment re-initiation provided the same criteria as above are met (2 consecutive negative MRD tests). Patients who are determined to have progressive disease per IMWG criteria (whether on treatment or observation schedule) will transition off study.
  Interventions: Drug: Elrantamab; Device: clonoSEQ

INTERVENTIONS:
Drug: Elrantamab — - Elranatamab will be dosed in 28-day cycles as follows:
  * C1D1: 12 mg SC priming dose
  * C1D3: 32 mg SC priming dose
  * C1D8, C1D15, C1D22: 76 mg SC
  * Cycle 2-Cycle 7: 76 mg SC on D1 and D15
  * Cycle 8 and subsequent cycles: 76 mg SC on D1
Device: clonoSEQ — FDA approved MRD testing

SUMMARY:
This study evaluates an individualized approach combining highly active maintenance treatment with elranatamab with peripheral blood-based clonotypic measurable residual disease (MRD) testing in patients with newly diagnosed multiple myeloma. The overall goal is to generate efficacy data for a personalized maintenance approach using bone marrow-based MRD testing (clonoSEQ) to guide post-autologous hematopoietic cell transplant (AHCT) maintenance with elranatamab for this patient population.

ELIGIBILITY:
Criteria for Pre-Screening Blood Draw

* Newly diagnosed multiple myeloma (either untreated or receiving first line therapy).
* Potentially eligible for autologous hematopoietic cell transplant (with or without tandem transplant) for frontline therapy.

Inclusion Criteria:

* At least 18 years of age
* Ability to understand and willingness to sign an IRB approved written informed consent document. (Legally authorized representatives may sign and give informed consent on behalf of study participants.)
* Received autologous hematopoietic cell transplantation (with or without tandem transplant) as part of frontline therapy for newly diagnosed IgG or IgA multiple myeloma. Frontline therapy in this setting is defined as treatment received prior to first relapse and may include multiple lines of therapy per the Rajkumar et al definition if treatment changes were made for either toxicity or inadequate response to initial induction.
* Received frontline treatment with at least a triplet regimen including a PI and an IMID (+/- an anti-CD38 antibody)
* Disease response of ≥ partial response (PR) by IMWG criteria at time of study screening (post-transplant).
* MRD-positive on Day 100 landmark assessment (80 to 160 days after AHCT), defined as >1 x 10-5 myeloma cells/cell by clonoSEQ assay (Adaptive Biotechnologies, Seattle, WA) performed on bone marrow aspirate.
* ECOG performance status ≤ 2
* All toxicities from prior treatment should have resolved to Grade ≤ 1 prior to enrollment.
* Adequate bone marrow and organ function within 28 days prior to start of treatment as defined below:

  * Platelets ≥ 75 k/cumm
  * Absolute neutrophil count ≥ 1.0 k/cumm
  * Hemoglobin ≥ 8 g/dL without the use of growth factors or transfusion for at least 2 weeks.
  * Total bilirubin ≤ 2 × upper limit of normal (ULN; ≤ 3 x ULN if documented Gilbert's syndrome)
  * Aspartate aminotransferase and alanine aminotransferase ≤ 2.5 × ULN
  * Creatinine clearance ≥ 30 ml/min.
* The effects of elranatamab on the developing human fetus are unknown. For this reason, women of childbearing potential and men must agree to use adequate contraception prior to study entry, for the duration of study participation, and for 5 months after end of treatment. Should a woman become pregnant or suspect she is pregnant while participating in this study, or should a man suspect he has fathered a child, s/he must inform her treating physician immediately.

Exclusion Criteria:

* Inability to identify a trackable clonoSEQ ID.
* A history of other malignancy with the exception of non-melanoma skin cancers, low or very low risk prostate cancer by NCCN criteria status post definitive therapy or currently on active surveillance, and malignancies for which all treatment was completed at least 2 years before registration and the patient has no evidence of disease. Adjuvant endocrine therapy for hormone receptor-positive breast cancer is not exclusionary.
* Currently receiving any other investigational agents.
* Prior BCMA-based treatment.
* CNS involvement of disease.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to elranatamab or other agents used in the study.
* Uncontrolled intercurrent illness including, but not limited to, plasma cell leukemia, POEMS syndrome, systemic amyloidosis, ongoing or active infection (bacterial, fungal, or viral).
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative serum pregnancy test within 28 days prior to first dose of elranatamab.
* HIV-infected if not on effective anti-retroviral therapy with undetectable viral load for 6 months. Patients with HIV who are receiving effective anti-retroviral therapy and have had an undetectable viral load for at least 6 months are eligible. HIV testing not required in the absence of known history of infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2024-12-20 (Actual); Primary Completion 2031-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Through completion of follow-up (up to 5 years)
  Progression-free survival (PFS) is defined as time to progression or death.
Proportion of patients achieving MRD negativity at the 10^-5 threshold per the clonoSEQ assay | Through completion of end of study visit (up to 36 months)

SECONDARY OUTCOMES:
Event-free survival (EFS) | Through completion of follow-up (up to 5 years)
  Composite of progression, death, or treatment intolerance (discontinuation due to toxicity)
Time to next therapy | Through completion of follow-up (up to 5 years)
  Time to next therapy (TTNT) is defined as the time to initiation of subsequent anti-myeloma therapy (excluding standard-of-care maintenance).
Maximum depth of response by IMWG criteria | Through completion of end of study visit (up to 36 months)
Proportion of patients achieving sustained MRD-negativity at the 10^-5 threshold per the clonoSEQ assay for at least 12 months | Through completion of end of study visit (up to 36 months)
  MRD negativity per the clonoSEQ assay will be defined as less than 1 myeloma cell per 10^6 bone marrow cells evaluated (i.e. <10-6)
Proportion of patients discontinuing therapy per MRD-guided protocol | Through completion of treatment (up to 36 months)
Time on treatment during study period | Through completion of treatment (up to 36 months)
Incidence and severity of treatment-related adverse events by CTCAE v5 | From start of treatment through 90 days after completion of treatment (up to 39 months)
Overall survival (OS) | Through completion of follow-up (up to 5 years)
  Overall survival (OS) is defined as time to death.
Proportion of patients resuming therapy per MRD-guided protocol | Through completion of treatment (up to 36 months)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Slade, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP
Access Criteria: Interested parties should contact the investigator to discuss access to de-identified datasets.

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu